CLINICAL TRIAL: NCT00414232
Title: Prospective Assessment of Symptoms and Quality of Life in Rectal Cancer Patients Receiving Chemo-Radiotherapy
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: J06109; NA_00004324 (Other: JHM IRB)
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Chemoradiation; Rectal Cancer receiving chemoradiation.
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective Assessment of Symptoms and Quality of Life in Rectal Cancer Patients Receiving Chemo-Radiotherapy.

DETAILED DESCRIPTION:
STUDY PLAN

1. Only the principal investigator, sub-investigators, and research nurse will be approaching potential participants. The above listed also will be the only consentors for the study. The recruitment process will occur during the outpatient visits being held at the Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins. HIPAA (Health Insurance Portability and Accountability Act ) and guidelines and good clinical practice will be followed at all times to ensure that the privacy of participants included in the recruitment process are strictly guarded.
2. Patients will be registered by the Radiation Oncology clinical subjects coordinator after eligibility is confirmed and informed consent is obtained.
3. The EORTC (European Organization for Research and Treatment of Cancer)QLQ- C30 (Quality of Life Questionnaire), QLQ-CR38 (Quality of Life Questionnaire), and QLQ-CR29 (Quality of Life Questionnaire) forms will be completed by patients at the following time point:

   1. Within 3 weeks prior to start of radiotherapy
   2. During the 4th week of radiotherapy (when treatment-related symptoms are expected to peak)
   3. Approximately one month after completion of radiotherapy during a follow-up visit
4. The QOL forms (QLC-C30, QLQ-CR38, and CR29) will be self-administered surveys. A nurse or other healthcare provider will be available to help the patient with any questions regarding the QOL forms.
5. The symptom inventory will be collected in an interview by a nurse or other healthcare provider at the following time points: d. Within 3 weeks prior to start of radiotherapy e. Once weekly during radiotherapy f. Approximately one month after completion of radiotherapy during a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* All of the following questions must be answered "yes" for a patient to be eligible for this protocol.

  1. Is there a working diagnosis of rectal cancer? YES NO
  2. Will the patient be receiving neoadjuvant concurrent chemotherapy and pelvic radiation? YES NO
  3. Is the pelvic radiation planned for a dose of 45-54 Gy and will it be delivered using a standard 3-field technique? YES NO
  4. Is the patient ≥ 18 years of age? YES NO
  5. Can the patient give informed consent? YES NO

Exclusion Criteria:

* All of the following questions must be answered "no" for a patient to be eligible for this protocol.

  1. Has there been prior radiation to the pelvis? YES NO
  2. Is the patient in the "special category" designated by the Public Health Service (patients younger than 18, pregnant women, and prisoners)? YES NO

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females greater than or equal to 18 years of age with a working diagnosis of rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) | 1 year
  Assessment of Quality of Life of Patients post standard of care radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Herman, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at The Johns Hopkins University, Baltimore, Maryland, United States